CLINICAL TRIAL: NCT00204607
Title: Induction of Specific Immune Responses Against Melanoma-Associated Antigens in Vivo by Intradermal Vaccination With Stabilized Tumor mRNA - a Clinical Phase I/II Trial
Brief Title: Intradermal Vaccination With Stabilized Tumor mRNA - a Clinical Phase I/II Trial in Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNA-Mel-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — RNA, Messenger

INTERVENTIONS:
Biological: mRNA
Drug: GM-CSF s.c.

SUMMARY:
vaccination protocol to induce specific immune responses against melanoma associated antigens by intradermal injections of mRNA coding for the corresponding antigen

DETAILED DESCRIPTION:
vaccination protocol to induce specific immune responses against melanoma associated antigens by intradermal injections of mRNA coding for the corresponding antigen. Antigens used are Melan-A, Mage-A1, Mage-A3, Survivin, GP100 and Tyrosinase. GM-CSF is used as an adjuvans. Phase I/II clinical trial to analyse safety and immune respones in stage III/IV melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* stage III/IV
* fresh frozen tumor-tissue
* age 18-75
* informed consent given
* Karnofsky >= 70%

Exclusion Criteria:

* systemic glucocorticoids
* brain metestasis
* other malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
toxicity
immune response

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof. Dr., Principal Investigator — University of Tuebingen, Department of dermatology
Locations (1):
- Department of Dermatology, University of Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Weide B, Pascolo S, Scheel B, Derhovanessian E, Pflugfelder A, Eigentler TK, Pawelec G, Hoerr I, Rammensee HG, Garbe C. Direct injection of protamine-protected mRNA: results of a phase 1/2 vaccination trial in metastatic melanoma patients. J Immunother. 2009 Jun;32(5):498-507. doi: 10.1097/CJI.0b013e3181a00068. PMID 19609242